CLINICAL TRIAL: NCT06443684
Title: Prospective, Observational Study of Molecular Residual, Dynamic Monitoring and Recurrence of Stage III Driver Mutated NSCLC
Brief Title: A Study of Molecular Residual, Dynamic Monitoring and Recurrence of Stage III Driver Mutated NSCLC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Lu Shun, Professor Chief of Shanghai Lung Cancer Center, Shanghai Chest Hospital
Other Study IDs: ADX-MRD-LC
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood samples processed into plasma, buffy coat,and serum Formalin-fixed paraffin-embedded tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Direct surgery: Stage III NSCLC eligible for direct surgery
  Interventions:
  Diagnostic Test: MRD（LC-10）include 10 lung cancer-related driver gene mutation site
  Interventions: Diagnostic Test: MRD
- Neoadjuvant and surgery: Stage III NSCLC eligible for neoadjuvant therapy followed by surgery
  Interventions:
  Diagnostic Test: MRD（LC-10）include 10 lung cancer-related driver gene mutation site
  Interventions: Diagnostic Test: MRD
- Chemoradiotherapy: Unresectable Stage III NSCLC eligible for Chemoradiotherapy.
  Interventions:
  Diagnostic Test: MRD（LC-10）include 10 lung cancer-related driver gene mutation site
  Interventions: Diagnostic Test: MRD

INTERVENTIONS:
Diagnostic Test: MRD — MRD（LC-10）include 10 lung cancer-related driver gene mutation site

SUMMARY:
The goal of this prospective, observational study is to explore the value of dynamic monitoring of minimal residual lesions in driver mutated stage III NSCLC for disease recurrence and prognosis assessment. The main question it aims to answer is:

1) Whether MRD(Minimal residual disease) status can predict recurrence events in stage III driven-mutant NSCLC in advance

DETAILED DESCRIPTION:
Non-small cell lung cancer in stage III (IIIa, IIIIb, IIIc) has a low survival rate, and the 5-year survival rate of stage III patients is less than 30%. In clinical studies of non-small cell lung cancer operable stage III driver gene mutations, postoperative targeted adjuvant therapy improves patient survival relative to postoperative chemotherapy.

The tumor patients still have residual malignant tumor cells in vivo during or after treatment, and minimal residual foci are released during cell necrosis or apoptosis. Early the domestic large lung cancer MRD((Minimal residual disease)) prospective research results, for the first time through the dynamic monitoring of MRD high negative predictive value defined the potential cure population, found that postoperative MRD negative population could not benefit from adjuvant therapy, clarify the existence of preoperative Non-shedding tumor does not affect postoperative MRD monitoring, and exploring the stage II / III MRD turn high risk of postoperative lung cancer. Therefore, for nearly 70% of patients with driver gene-positive non-small-cell lung cancer, detecting clear driver gene mutations in the peripheral blood is expected to stratify the risk of recurrence/progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage III non-small cell lung cancer were confirmed by imaging and histological biopsy
2. Age≥ 18
3. ECOG PS:0-1
4. Tumor molecular testing by EBUS or biopsy confirmed positive for one or more of the following driver genes:EGFR\ALK\ROS1\RET\KRAS\PIK3CA\BRAF\HER2\MET
5. Patients who met and agreed to surgery or radical chemoradiotherapy, and the remaining samples after cutting tissue sections did not affect the possible further clinical treatment of the subject
6. Provide 20 mL peripheral blood samples periodically
7. The subjects volunteered to join the study, and signed the informed consent form, with good compliance, and actively cooperated with the hospital for routine clinical diagnosis and treatment follow-up

Exclusion Criteria:

1. Patients with other malignancies within 5 years
2. According to the investigator, the patient also had other diseases that may affect the follow-up and short-term survival
3. The subject had other factors that may lead to the termination of the study, such as other serious diseases (including mental illness), serious laboratory abnormalities, and family or social factors that affected the safety of the subject, or the collection of data and samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 305 The main research purpose of this project is to associate the MRD status of driver gene positive patients with 12 months of recurrent events. The follow-up is 2 years, so according to the number of patients with stage IIIA NSCLC in each center, and the patient enrollment is planned within 1 year. A total of 305 stage III NSCLC patients were collected
Sampling Method: Non-Probability Sample
Enrollment: 305 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of MRD status in driver gene-positive NSCLC patients with 12-month relapse events | 2022.12--2025.03
  Patients are defined as MRD positive if lung cancer driver genes are detected in peripheral blood post-surgery using NGS methods, and radiological recurrence is based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Correlation of MRD status in driver gene-positive NSCLC patients with RFS | 2022.12--2025.03
  Patients are defined as MRD positive if lung cancer driver genes are detected in peripheral blood post-surgery using NGS methods, and radiological recurrence is based on RECIST 1.1 criteria.
Correlation of MRD status in driver gene-positive NSCLC patients with OS | 2022.12--2025.03
  Patients are defined as MRD positive if the NGS method detects lung cancer driver gene positivity in the peripheral blood post-surgery.
Correlation of MRD status in driver gene-positive NSCLC patients with 24-month relapse events | 2022.12--2025.03
  Patients are defined as MRD positive if lung cancer driver genes are detected in peripheral blood post-surgery using NGS methods, and radiological recurrence is based on RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, M.D., Principal Investigator — Shanghai Chest Hospital
Locations (11):
- China (11):
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Chest hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No